CLINICAL TRIAL: NCT02138890
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Pilot Study of a Single, Intra-Articular Injection of Autologous Protein Solution (APS) in Patients With Osteoarthritis (OA) of the Knee
Brief Title: APSS-33-00: A Multicenter, Pilot Study of Autologous Protein Solution (APS) in Knee Osteoarthritis (OA)
Acronym: PROGRESS II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BBI.CR.APS1.14
Record Dates: First submitted 2014-05-01; First posted 2014-05-15 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-01

CONDITIONS: Osteoarthritis, Knee
Keywords: Autologous Protein Solution; APS; Osteoarthritis; Intra Articular Injection
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APS injection (Experimental): Autologous Protein Solution
  Interventions: Device: APS
- Control (Placebo Comparator): Saline
  Interventions: Device: Saline

INTERVENTIONS:
Device: APS — Intra-articular Injection
  Arms: APS injection
Device: Saline — Intra-articular injection
  Arms: Control

SUMMARY:
This double-blind, multicenter, randomized, controlled trial (RCT) will evaluate the efficacy of a single dose of Autologous Protein Solution (APS) in patients with osteoarthritis (OA) of the knee who have failed at least 1 conservative osteoarthritis (OA) therapy (e.g. physiotherapy, simple analgesics, intra-articular injection).

DETAILED DESCRIPTION:
A double-blind, multicenter, randomized, controlled trial (RCT) that will evaluate the efficacy of a single dose of Autologous Protein Solution (APS) in patients with Osteoarthritis (OA) of the knee who have failed at least 1 conservative OA therapy (e.g. physiotherapy, simple analgesics, intra-articular injection).

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥40 years and ≤75 years.
* Willingness and ability to comply with the study procedures and visit schedules and ability to follow verbal and written instructions.
* Diagnosis of knee osteoarthritis (OA) Grade 2 or 3 according to the Kellgren-Lawrence scale
* Body mass index (BMI) ≤ 40.
* Failed at least 1 conservative OA therapy
* Signed an independent ethics committee (IEC) approved informed consent form (ICF).

Main Exclusion Criteria:

* Intra-articular Hyaluronic (HA) injection within 6 months- On Day 1 (pre-injection), presence of active infection or abnormal effusion in the knee as noted by a physical examination (e.g., erythema, redness, heat, swelling).
* Presence of symptomatic OA in the non-study knee.
* Diagnosed with rheumatoid arthritis (RA), Reiter's syndrome, psoriatic arthritis, ankylosing spondylitis, chondromalacia, arthritis secondary to other inflammatory diseases (e.g., inflammatory bowel disease [IBD], sarcoidosis, or amyloidosis) or of metabolic origin.
* Diagnosis of isolated patella-femoral joint osteoarthritis.
* Valgus/varus deformity judged by the investigator to be clinically significant.
* Disease of spine, hip or other lower extremity joints of sufficient degree to affect assessment of the signal knee. Patients with TKR at the contra-lateral knee or THR in either hip may be enrolled provided sufficient pain relief after TKR or THR which does not require additional analgesic relief.
* Untreated acute traumatic injury of the index knee.
* Presence of a symptomatic meniscal tear in the index knee
* Limited daily activity for reasons other than OA.
* Presence of surgical hardware or other foreign body in the index knee.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-05; Primary Completion 2015-10 (Actual); Study Completion 2020-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: DiMartino, MD, Principal Investigator — Bologna (Italy)
Locations (4):
- Krems Hospital, Krems, Austria
- Monica Hospitals, Antwerp, Belgium
- Rizzoli Orthopaedic Institute, Bologna, Italy
- Oslo University, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kon E, Engebretsen L, Verdonk P, Nehrer S, Filardo G. Autologous Protein Solution Injections for the Treatment of Knee Osteoarthritis: 3-Year Results. Am J Sports Med. 2020 Sep;48(11):2703-2710. doi: 10.1177/0363546520944891. PMID 32870042
- [Derived] Kon E, Engebretsen L, Verdonk P, Nehrer S, Filardo G. Clinical Outcomes of Knee Osteoarthritis Treated With an Autologous Protein Solution Injection: A 1-Year Pilot Double-Blinded Randomized Controlled Trial. Am J Sports Med. 2018 Jan;46(1):171-180. doi: 10.1177/0363546517732734. Epub 2017 Oct 10. PMID 29016185

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multicenter study, with 4 centers in Belgium, Italy, Austria and Norway. The first subject was enrolled on 8 May 2014.
Period: Overall Study
Arm/Group | APS Injection | Control
Started (Subjects were followed up for 12 months and if they consent, for a long term follow-up of 5 years.) | 31 | 15
Completed | 30 | 15
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Patients who have OA in the knee who have failed at least 1 prior conservative OA therapy (e.g. physiotherapy, simple analgesics, intra-articular injection).
Groups:
- APS Injection: Autologous Protein Solution (APS): Intra-articular Injection
- Total: Total of all reporting groups
Arm/Group | APS Injection | Control | Total
Number analyzed (Participants) | 31 | 15 | 46
Age, Continuous [Mean (Full Range); unit: years] | 57.4 [41 to 68] | 54.1 [44 to 67] | 55.8 [41 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 19
  Male | 18 | 9 | 27
Region of Enrollment [Number; unit: participants]
  Belgium | 5 | 3 | 8
  Norway | 14 | 6 | 20
  Italy | 12 | 6 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 6 Months in Pain Measured With WOMAC Questionnaire (Day 1, Week 2, Month 1, 3 and 6)
Description: The WOMAC LK 3.1 questionnaire is a validated tool commonly used for assessing knee pain, stiffness, and function. The WOMAC LK 3.1 questionnaire has 24 items that the patient addresses about the knee: 5 items on the pain subscale, 2 on the stiffness subscale, and 17 on the physical function subscale. Each item is answered on a 5-point Likert scale, with grading from 0 (none or never) to 4 (extreme or always). A higher score indicates worse pain, stiffness, or functional limitation.
  The WOMAC pain subscale consisted of five questions scored from 0 to 4. The pain has a range of 0 (no pain) to 20 (maximal pain).
Time Frame: 6 months
Population: The safety/ITT population analysis population was utilized for this analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- APS Injection: Autologous Protein Solution: Intra-articular Injection
Arm/Group | APS Injection | Control
Number analyzed (Participants) | 31 | 15
scores on a scale
  Day 1 | 11.5 (2.4) | 11.8 (1.9)
  Week 2 | 8.6 (4.0) | 8.7 (4.1)
  1 Months | 7.0 (4.1) | 8.4 (3.4)
  3 Months | 5.6 (3.9) | 5.7 (4.2)
  6 Months | 5.0 (3.8) | 5.6 (4.1)

2. Primary Outcome: Pain Measured With WOMAC Questionnaire Subscale Pain at Day 1, Week 2, 1 Month, 3 Months, 6 Months and 12 Months.
Description: as for outcome 1
Time Frame: 12 Months
Population: This data describes mITT/PP analysis set
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | APS Injection | Control
Number analyzed (Participants) | 29 | 14
scores on a scale
  Day 1 | 11.5 (2.4) | 11.8 (1.9)
  Week 2 | 8.6 (4.0) | 8.7 (4.1)
  1 Month | 7.0 (4.1) | 8.4 (3.4)
  3 Months | 5.6 (3.9) | 5.7 (4.2)
  6 Months | 5.0 (3.8) | 5.6 (4.1)
  12 Months | 4.3 (4.0) | 6.3 (3.9)

3. Secondary Outcome: Pain Measured With Visual Analogue Scale at Day 1, Week 2, 1 Month, 3 Months, 6 Months and 12 Months
Description: The Visual Analogue Scale is a common tool for measuring general pain. A 100 mm line is marked from 0 to 10 in 10 mm increments. Knee pain severity is indicated by drawing a vertical mark at the point on the line that best represents the severity of pain. No pain is indicated by the 0 at the far left, and the worst possible pain is indicated by the 100 at the far right.
Time Frame: 12 Months
Population: The 12 Month efficacy analyses were done on the mITT/PP analysis set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | APS Injection | Control
Number analyzed (Participants) | 29 | 14
scores on a scale
  Day 1 | 5.5 (2.2) | 6.5 (1.8)
  Week 2 | 4.7 (2.6) | 5.3 (2.0)
  1 Month | 4.0 (2.3) | 5.2 (2.1)
  3 Months | 3.3 (2.0) | 3.9 (2.1)
  6 Months | 3.1 (2.5) | 4.1 (2.3)
  12 Months | 2.6 (2.5) | 4.8 (2.2)

4. Secondary Outcome: Stiffness Measured With WOMAC Subscale Stiffness Questionnaire at Day 1, Week 2, 1 Month, 3 Months, 6 Months and 12 Months
Description: The WOMAC LK 3.1 questionnaire is a validated tool commonly used for assessing knee pain, stiffness, and function. The WOMAC LK 3.1 questionnaire has 24 items that the patient addresses about the knee: 5 items on the pain subscale, 2 on the stiffness subscale, and 17 on the physical function subscale. Each item is answered on a 5-point Likert scale, with grading from 0 (none or never) to 4 (extreme or always). A higher score indicates worse pain, stiffness, or functional limitation.
  The WOMAC Stiffness subscale consisted of two questions scored from 0 to 4. The Stiffness has a range of 0(no stiffness) to 8 (maximal stiffness)
Time Frame: 12 months
Population: The 12 Month efficacy analyses were done on the mITT/PP analysis set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | APS Injection | Control
Number analyzed (Participants) | 29 | 14
scores on a scale
  Day 1 | 4.8 (1.7) | 5.0 (1.2)
  Week 2 | 4.0 (2.0) | 3.6 (1.6)
  1 Month | 3.3 (1.8) | 3.9 (1.3)
  3 Months | 3.0 (1.6) | 3.4 (1.5)
  6 Months | 2.7 (2.0) | 2.9 (1.6)
  Month 12 | 2.7 (1.7) | 3.0 (2.0)

5. Secondary Outcome: Function on Daily Living Measured With WOMAC Subscale Questionnaire Physical Functioning at Day 1, Week 2, 1 Month, 3 Months, 6 Months and 12 Months
Description: The WOMAC LK 3.1 questionnaire is a validated tool commonly used for assessing knee pain, stiffness, and function. The WOMAC LK 3.1 questionnaire has 24 items that the patient addresses about the knee: 5 items on the pain subscale, 2 on the stiffness subscale, and 17 on the physical function subscale. Each item is answered on a 5-point Likert scale, with grading from 0 (none or never) to 4 (extreme or always). A higher score indicates worse pain, stiffness, or functional limitation.
  The WOMAC Physical Functioning subscale consisted of seventeen questions scored from 0 to 4. The Physical Functioning has a range of 0 (no functional limitation) to 68 (maximal functional limitation)
Time Frame: 12 months
Population: The 12 Month efficacy analyses were done on the mITT/PP analysis set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | APS Injection | Control
Number analyzed (Participants) | 29 | 14
scores on a scale
  Day 1 | 34.9 (12.4) | 38.1 (9.3)
  Week 2 | 30.2 (14.8) | 29.4 (15.1)
  1 Month | 24.9 (14.7) | 28.9 (10.8)
  3 Months | 21.5 (14.5) | 20.4 (13.4)
  6 Months | 18.5 (13.0) | 18.0 (12.7)
  Month 12 | 15.6 (13.8) | 20.4 (12.3)

6. Secondary Outcome: Pain as Measured With Knee Injury and Osteoarthritis Outcome Score (KOOS) Subscale Pain at Day 1, Week 2, 1 Month, 3 Months, 6 Months and 12 Months
Description: The KOOS questionnaire is a commonly used instrument to assess the patient's opinion about their knee and associated problems. KOOS consists of 5 subscales: Pain (9 questions), Symptoms (7 questions), Function in daily living (ADL) (17 questions), Function in sport and recreation (Sport/Rec) (5 questions) and knee related Quality of Life (QOL) (4 questions). The previous week is used as the time period for answering the questions.
  A higher score on the KOOS questionnaire indicates no problems, and 0 indicates extreme problems. Each subscale score is calculated independently. The mean score of the individual items of each subscale is calculated and divided by 4 (the highest possible score for a single answer option). on). Traditionally in orthopedics, 100 indicates no problems and 0 indicates extreme problems. The normalized score is transformed to meet this standard.
Time Frame: 12 months
Population: The 12 Month efficacy analyses were done on the mITT/PP analysis set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | APS Injection | Control
Number analyzed (Participants) | 29 | 14
scores on a scale
  Day 1 | 39.9 (13.1) | 37.9 (10.1)
  Week 2 | 51.1 (19.7) | 48.0 (16.6)
  1 Month | 58.2 (19.5) | 51.8 (16.3)
  3 Months | 64.1 (20.7) | 64.7 (20.8)
  6 Months | 66.6 (20.3) | 65.9 (19.2)
  Month 12 | 70.6 (21.5) | 61.1 (18.5)

7. Secondary Outcome: Symptoms Measured With Knee Injury and Osteoarthritis Outcome Score (KOOS) Subscale Symptoms at Day 1, Week 2, 1 Month, 3 Months, 6 Months and 12 Months
Description: as for outcome 6
Time Frame: 12 months
Population: The 12 Month efficacy analyses were done on the mITT/PP analysis set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | APS Injection | Control
Number analyzed (Participants) | 29 | 14
scores on a scale
  Day 1 | 47.8 (19.3) | 46.4 (12.1)
  2 Weeks | 55.4 (22.0) | 54.9 (17.1)
  1 Month | 64.2 (20.4) | 56.1 (15.3)
  3 Months | 65.3 (17.4) | 62.5 (14.6)
  6 Months | 67.2 (20.3) | 63.3 (15.1)
  Month 12 | 68.4 (21.4) | 58.2 (17.4)

8. Secondary Outcome: Function in Daily Living Measured With Knee Injury and Osteoarthritis Outcome Score (KOOS) Subscale Function in Daily Living at Day 1, Week 2, 1 Month, 3 Months, 6 Months and 12 Months
Description: as for outcome 6
Time Frame: 12 months
Population: The 12 Month efficacy analyses were done on the mITT/PP analysis set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | APS Injection | Control
Number analyzed (Participants) | 29 | 14
scores on a scale
  Day 1 | 48.6 (18.3) | 44.0 (13.7)
  Week 2 | 55.5 (21.8) | 56.8 (22.2)
  1 Month | 63.4 (21.6) | 57.5 (15.9)
  3 Months | 68.3 (21.3) | 70.0 (19.8)
  6 Months | 72.8 (19.1) | 73.5 (18.7)
  Month 12 | 77.0 (20.3) | 70.0 (18.1)

9. Secondary Outcome: Sports and Recreational (Sport/Rec) Activities Measured With Knee Injury and Osteoarthritis Outcome Score (KOOS) Subscale Sport/Rec at Day 1, Week 2, 1 Month, 3 Months, 6 Months and 12 Months
Description: as for outcome 6
Time Frame: 12 months
Population: The 12 Month efficacy analyses were done on the mITT/PP analysis set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | APS Injection | Control
Number analyzed (Participants) | 29 | 14
scores on a scale
  Day 1 | 23.1 (25) | 14.3 (9.4)
  Week 2 | 29.0 (22.4) | 23.2 (15.3)
  1 Month | 30.7 (27.6) | 26.6 (18.8)
  3 Months | 37.7 (27.1) | 40.2 (25.1)
  6 Months | 39.1 (25.3) | 42.1 (23.7)
  Month 12 | 47.1 (29.5) | 37.1 (27.9)

10. Secondary Outcome: Quality of Life Measured With Knee Injury and Osteoarthritis Outcome Score (KOOS) Subscale Quality of Life Questionnaire at Day 1, Week 2, 1 Month, 3 Months, 6 Months and 12 Months
Description: as for outcome 6
Time Frame: 12 months
Population: The 12 Month efficacy analyses were done on the mITT/PP analysis set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | APS Injection | Control
Number analyzed (Participants) | 29 | 14
score on a scale
  Day 1 | 26.5 (13.8) | 22.3 (8.7)
  Week 2 | 29.0 (22.4) | 23.2 (15.3)
  1 Month | 30.7 (27.6) | 26.8 (18.8)
  3 Months | 37.7 (27.1) | 40.2 (25.1)
  6 Months | 39.1 (25.3) | 42.1 (23.7)
  Month 12 | 51.3 (25.3) | 38.4 (19.3)

11. Secondary Outcome: Physical Functioning Measured With Short Form-36 (SF-36) Subscale Physical Functioning Questionnaire at Day 1, 6 Months and 12 Months
Description: The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. Eight subscales of the Short Form-36 questionnaire are used to derive Physical Component and Mental Component measures
Time Frame: 12 Months
Population: The 12 Month efficacy analyses were done on the mITT/PP analysis set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | APS Injection | Control
Number analyzed (Participants) | 29 | 14
score on a scale
  Day 1 | 35.8 (10.0) | 33.9 (9.4)
  6 Months | 43.3 (9.2) | 42.0 (9.6)
  Month 12 | 43.5 (10.2) | 42.2 (10.2)

12. Secondary Outcome: Mental Health Measured With Short Form-36 (SF-36) Subscale Mental Health Questionnaire at Day 1, 6 Months and 12 Months
Description: The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: 12 Months
Population: The 12 Month efficacy analyses were done on the mITT/PP analysis set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | APS Injection | Control
Number analyzed (Participants) | 29 | 14
scores on a scale
  Day 1 | 51.5 (8.5) | 50.8 (8.9)
  Month 6 | 54.1 (7.7) | 53.8 (6.0)
  Month 12 | 55.2 (7.4) | 53.0 (7.9)

13. Secondary Outcome: Role Physical Measured With Short Form-36 (SF-36) Subscale Role Physical Questionnaire at Day 1, 6 Months and 12 Months
Description: as for outcome 12
Time Frame: 12 Months
Population: The 12 Month efficacy analyses were done on the mITT/PP analysis set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | APS Injection | Control
Number analyzed (Participants) | 29 | 14
scores on a scale
  Day 1 | 38.5 (12.0) | 38.8 (10.4)
  Month 6 | 44.1 (12.4) | 45.7 (11.1)
  Month 12 | 46.0 (10.9) | 42.4 (9.3)

14. Secondary Outcome: Bodily Pain Measured With Short Form-36 (SF-36) Subscale Bodily Pain Questionnaire at Day 1, 6 Months and 12 Months
Description: as for outcome 12
Time Frame: 12 Months
Population: The 12 Month efficacy analyses were done on the mITT/PP analysis set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | APS Injection | Control
Number analyzed (Participants) | 29 | 14
scores on a scale
  Day 1 | 36.7 (7.6) | 35.0 (7.9)
  Month 6 | 44.0 (10.9) | 43.7 (7.2)
  Month 12 | 47.0 (9.3) | 39.2 (7.0)

15. Secondary Outcome: General Health Measured With Short Form-36 (SF-36) Subscale General Health Questionnaire at Day 1, 6 Months and 12 Months
Description: as for outcome 12
Time Frame: 12 Months
Population: The 12 Month efficacy analyses were done on the mITT/PP analysis set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | APS Injection | Control
Number analyzed (Participants) | 29 | 14
scores on a scale
  Day 1 | 36.7 (7.6) | 35.0 (7.9)
  Month 6 | 44.0 (10.9) | 43.7 (7.2)
  Month 12 | 47.0 (9.3) | 39.2 (7.0)

16. Secondary Outcome: Vitality Measured With Short Form-36 (SF-36) Subscale Vitality Questionnaire at Day 1, 6 Months and 12 Months
Description: as for outcome 12
Time Frame: 12 Months
Population: The 12 Month efficacy analyses were done on the mITT/PP analysis set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | APS Injection | Control
Number analyzed (Participants) | 29 | 14
scores on a scale
  Day 1 | 51.7 (9.9) | 50.6 (7.6)
  Month 6 | 54.0 (8.8) | 52.4 (6.5)
  Month 12 | 54.6 (9.9) | 53.1 (6.2)

17. Secondary Outcome: Social Functioning Measured With Short Form-36 (SF-36) Subscale Social Functioning Questionnaire at Day 1, 6 Months and 12 Months
Description: as for outcome 12
Time Frame: 12 Months
Population: The 12 Month efficacy analyses were done on the mITT/PP analysis set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | APS Injection | Control
Number analyzed (Participants) | 29 | 14
scores on a scale
  Day 1 | 43.7 (10.9) | 44.5 (10.8)
  Month 6 | 49.6 (9.7) | 51.4 (7.4)
  Month 12 | 51.5 (8.3) | 47.6 (9.7)

18. Secondary Outcome: Role Emotional Measured With Short Form-36 (SF-36) Subscale Role Emotional Questionnaire at Day 1, 6 Months and 12 Months
Description: as for outcome 12
Time Frame: 12 Months
Population: The 12 Month efficacy analyses were done on the mITT/PP analysis set.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | APS Injection | Control
Number analyzed (Participants) | 29 | 14
scores on a scale
  Day 1 | 44.0 (13.7) | 39.5 (13.5)
  Month 6 | 48.1 (10.7) | 47.5 (10.4)
  Month 12 | 49.6 (10.5) | 42.5 (9.8)

ADVERSE EVENTS:
Time Frame: Day 1, week 2, month 1, month 3, month 6 and month 12
Description: Adverse Event reporting through 12-Month time point
Arm/Group | APS Injection | Control
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/31 | 1/15
Other Adverse Events (participants affected / at risk) | 14/31 | 6/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APS Injection (N=31) | Control (N=15)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Meniscus Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APS Injection (N=31) | Control (N=15)
Toothache (Gastrointestinal disorders) | 2 (4) | 0 (0)
Pain (General disorders) | 1 (2) | 0 (0)
cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vitamine D Deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (7)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 1 (1)
Alcoholic hangover (Psychiatric disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
pyrexia (General disorders) | 0 (0) | 1 (1)
influenza like ilness (General disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (8) | 1 (1)
Joint crepitation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint warmth (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Rheumatic disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less